CLINICAL TRIAL: NCT03391024
Title: Non-Contact Intraoperative Optical Imaging During Instrumentation Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Victor Yang, Senior Scientist, Physical Sciences Platform, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 177-2013
Record Dates: First submitted 2017-12-18; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Computer-assisted Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBL Experimental Navigation System (Experimental): As this is a single arm trial, all participants receive treatment.
  Interventions: Device: BBL Experimental Navigation System

INTERVENTIONS:
Device: BBL Experimental Navigation System — Comparison of accuracy of screw placement using experimental system while navigated with clinically approved system.

SUMMARY:
For a significant number of patients suffering from back pain, even basic daily activities become impossible. It is at this time that spinal surgery becomes necessary in order to improve the patient's quality of life. To combat these symptoms, surgical implants (e.g. pedicle screws, rods, etc.) are used to aid in stabilizing and correcting the deformities of the spine, particularly after spinal decompression. Surgical navigation has a great potential to improve the accuracy of correctly implanting these devices; however, present technologies rely on intraoperative imaging that uses ionizing radiation (e.g. computed tomography, fluoroscopy, etc.), require cumbersome set-ups, the physical attachment of fiducial markers, and cannot account for patient motion. Therefore, the investigators propose a real-time intraoperative optical topographical imaging based surgical guidance system capable of accurately guiding the placement of implanted devices such as pedicle screws.

DETAILED DESCRIPTION:
The hypothesis is that optical visualization of surgically exposed bony anatomy with computerized navigation can accurately estimate subsurface anatomy and in the future, potentially guide the placement of pedicle screws during spinal surgery. The specific research aims are as follows: i) an intraoperative non-contact optical imaging system can quantify the entry point and trajectory of pedicle screws implanted by the spine surgeon; and ii) intraoperative optical imaging can predict the entry point and trajectory of pedicle screws as verified by post-operative computed tomography (CT) scans.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Able to provide consent, or have substitute decision maker available FOR SPINAL INDICATIONS
* Scheduled to undergo spinal instrumentation surgery involving pedicle screw insertion
* Scheduled for pre-operative CT scan and the surgical plan includes open exposure of the posterior bony elements of one or more level(s) of the vertebra(e)
* No contra-indication for a post-operative CT scan FOR CRANIAL INDICATIONS
* scheduled to undergo cranial surgery
* Scheduled for pre-operative CT or MRI scan
* No contra-indication for post-operative CT scan

Exclusion Criteria:

* Previous spinal decompression with significant laminectomy performed at the level intended for instrumentation
* Previous spinal decompression with laminoplasty performed at the level intended for instrumentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
Pilot hole and screw trajectory accuracy as compared between post-operative CT and intraoperative images | Within 1 week of screw placement
  Comparison and quantification of accuracy of pilot holes including entry point and trajectory as taken from experimental navigation system as compared to absolute (or actual) entry point and trajectory of screws as determined by post-operative computed tomography scans.

CONTACTS AND LOCATIONS:
Overall Officials: Victor XD Yang, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merloz P, Tonetti J, Eld A, et al, Computer-assisted versus manual spine surgery: Clinical report, Springer Berlin, 1997.
- [Background] Rampersaud YR, Simon DA, Foley KT. Accuracy requirements for image-guided spinal pedicle screw placement. Spine (Phila Pa 1976). 2001 Feb 15;26(4):352-9. doi: 10.1097/00007632-200102150-00010. PMID 11224881
- [Background] Zdichavsky M, Blauth M, Knop C, Graessner M, Herrmann H, Krettek C, Bastian L, Accuracy of Pedicle Screw Placement in Thoracic Spine Fractures, European Journal of Trauma, 30:234-240, 2004